CLINICAL TRIAL: NCT04877509
Title: Micronutrient Status Involved in Immunity in Elderly Patients With COVID-19
Acronym: MicroCovAging
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL20_0730 A067
Record Dates: First submitted 2021-03-04; First posted 2021-05-07 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-03

CONDITIONS: Covid19
Keywords: Covid19; Micronutriments; Elderly
MeSH Terms: conditions — COVID-19 | interventions — Selenium; Zinc; Copper; Vitamin A; Fumigant 93

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Over 50 year's COVID-19 patients hospitalized at HCL from 1st March to 29th May 2020.
  Interventions: Biological: Selenium, Zinc and Copper, Vitamin A, D, E plasma concentrations during patient hospitalization

INTERVENTIONS:
Biological: Selenium, Zinc and Copper, Vitamin A, D, E plasma concentrations during patient hospitalization — Micronutrient assays on heparinized plasma.

SUMMARY:
During the ongoing COVID-19 pandemic, age was clearly the major factor of mortality. Increasing age was strongly associated with this risk, with the upper 80 years age group having more than 12-fold increased risk compared with those aged 50-59 years. Male gender was also associated with a doubling of risk.

The elderly subject is particularly exposed to global denutrition with risk of micronutrients deficiencies such as vitamins and trace elements. Those deficits expose to lower immunity. In addition, viral infection as COVID-19 can also worsen these deficits.

In general, low levels or intakes of micronutrients such as Zn, Se and vitamin A have been associated with adverse clinical outcomes during viral infections. This notion has been confirmed in a recent review proposing that besides vitamins A and D also B vitamins, vitamin C, omega-3 polyunsaturated fatty acids, as well as selenium, zinc and iron should be considered in the assessment of micronutrients in COVID-19 patients.

In this context, the MicroCovAging study will evaluate copper, zinc and selenium, vitamin A, D and E status in elderly subjects affected by COVID- 19 and to correlate this status with prognosis of this disease.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized adult patient ≥ 50 years at the time of admission,
* Suffering from confirmed COVID-19 (positive quantitative PCR for SARS-CoV-2 and/or chest scanner suggestive of COVID-19),
* Informed and non-opposed to the research. Patient will be informed of the study by his medical doctor during hospitalization or by post thanks to a generic information sheet dedicated to COVID-19 researches.

Exclusion Criteria:

* Adult patient < 50 years at the time of admission
* Negative quantitative PCR for SARS-Cov-2

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is an observational study based on a monocentric historical cohort of ≥ 50 years patients hospitalized at HCL from 1st March 2020 to 30th May 2020and suffering from COVID-19.
Sampling Method: Non-Probability Sample
Enrollment: 229 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Selenium, Zinc and Copper, Vitamin A, D and E plasma concentrations of 229 over 50 year's patients hospitalized suffering from COVID-19. | Up to 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Chls Cbap, Pierre-Bénite, France

REFERENCES:
- See also: Related Info — https://www.medrxiv.org/content/10.1101/2020.05.06.20092999v1